CLINICAL TRIAL: NCT06885112
Title: Clinical Study to Evaluate the Improvement in Hair Loss in Skin of Color Treated With Fractional Non-Ablative Laser
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-FoLix-24-01
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-03

CONDITIONS: Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- healthy subjects with moderate hair loss stage and skin color type 5 or 6 (Experimental): The FoLix is FDA cleared for hair loss treatments in patients with skin type 1 to 4. It is no being studied for patients with skin type 5 and 6 to allow expending the product labeling
  Interventions: Device: FoLix treatment for improving the scalp hair appearance

INTERVENTIONS:
Device: FoLix treatment for improving the scalp hair appearance — The study patients will receive 4 FoLix treatment in 4 weeks intervals. the scalp hair improvement will be evaluated by 3 blinded assessors who shall review before and after images, as well as hair count data

SUMMARY:
The study incudes 18 to 55 y/o healthy subjects with moderate hair loss stage and Fitzpatrick skin type 5 or 6

DETAILED DESCRIPTION:
The FoLix laser system contains Erbium:Glass Fiber Laser Technology with a wavelength of 1565 nm. It is the first FDA cleared fractional laser device for treatment of hair loss that has demonstrated safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male and females between 21 - 55 years of age, inclusive.
* Have Fitzpatrick Skin Type V to VI.
* Have mild to moderate hair loss (Ludwig scale I-II for women, Norwood-Hamilton scale I-III for males)
* Have self-reported thinning or hair loss for more than 6 months prior to screening but less than 5 years.
* Clinically confirmed to have hair loss or thinning by the investigator via physical exam
* Didn't receive hair-loss treatments or participated in a clinical study using 1565 NAFL device
* In good general health, as determined by the Investigator
* Willing and able to attend all study visits
* Willing to maintain the same hair style as at the Screening Visit for the duration of the study. If coloring hair, willing to color it with the same frequency of usage as in the past, making sure not to color within 1-week before and 1-week after an in-office appointment
* Willing to use a mild non-medicated shampoo and conditioner for the duration of the study (medicated shampoo and conditioner refer to any prescription shampoo or conditioner as well as any over-the counter medicated shampoo or conditioner, such as those for treatment of dandruff or promoting hair growth)
* Have a negative urine pregnancy test at screening and be using, and continue to use for the duration of the study, an effective contraception method (i.e., abstinence, barrier control, intrauterine device [IUD], or hormonal [estrogen/progestin] contraceptives) for at least one menstrual cycle prior to study; if using IUD or hormonal contraceptives - then at least 2 years prior to screening, the initiation of which should not have been associated with initiation of hair loss/thinning.
* Be willing and able to cooperate with the requirements of the study including images taken using a smart camera (multi-spectral) of several skin conditions
* Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board
* Be able to complete and understand the various rating instruments in English
* Sponsor approved global image assessment of degree of thinning / hair loss

Exclusion Criteria:

* Clinical diagnosis of alopecia areata or scarring forms of alopecia
* Patient is of skin type I-IV
* Scalp hair loss on the treatment area, due to disease, injury, or medical therapy
* Subjects who are pregnant, planning to become pregnant or breastfeeding. A urine pregnancy test will be done to rule out pregnancy. Subjects of childbearing potential who are not using an approved method of birth control (oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence). Females of non-childbearing potential are defined as postmenopausal (e.g.: absence of menstrual bleeding for one year), hysterectomy or bilateral oophorectomy
* Current skin disease (e.g., psoriasis, atopic dermatitis, skin cancer, eczema, sun damage, seborrheic dermatitis), cuts and or abrasions on the scalp or condition (e.g., sunburn, tattoos) on the treatment area that, in the opinion of the Investigator, might put the subject at risk or interfere with the study conduct or evaluations
* Participated in a previous 1565 NAFL study or treatment
* History of surgical correction of hair loss on the scalp/ Hair transplants.
* Use of any products or devices purported to promote scalp hair growth (e.g., finasteride or minoxidil) within the 90 days prior to the Baseline Visit.
* Use of anti-androgenic therapies (e.g., spironolactone, flutamide, cyproterone acetate, cimetidine) within 60 days prior to the Baseline Visit.
* No history of burning, flaking, itching, and stinging of the scalp.
* A chronic condition of high severity dandruff.
* History of malignancy (except scc and bcc skin cancers) or undergoing chemotherapy or radiation treatments.
* A known history of autoimmune thyroid disease, any other thyroid disorder/abnormality or other autoimmune disorders that in the opinion of the investigator may interfere with the study treatment.
* A known history of untreated or uncontrolled depression or bipolar disease or any other condition that may impact the subject's participation.
* Recent utilization of low level lasers for treating hair loss (past 6 months).
* Has any condition that the treating investigator or PI thinks may put the Subject at risk or interfere with their participation in the study.
* Is involved in any injury litigation claims.
* Known history or recent bloodwork indicating iron deficiency (ferritin level is less than 30 ng/mL), bleeding disorders or platelet dysfunction syndrome as well as subjects receiving anticoagulant therapy or smokers with usage >20 cigarettes/day.
* Use of any medications that are known to potentially cause hair loss or affect hair growth, as determined by PI.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-02-21 (Estimated); Study Completion 2027-02-21 (Estimated)

PRIMARY OUTCOMES:
improvement in scalp hair appearance by comparing before and after images | 12 months
  The primary endpoint, the proportion of picture sets correctly classified as before/after by at least 2 of the 3 blinded reviewers, will be summarized by a count a percentage with exact two-sided 95% confidence interval. If the lower limit is greater than 70%, the null hypothesis will be rejected, and the endpoint will be deemed successfully met.
  There will be no formal interim statistical analysis.

SECONDARY OUTCOMES:
Hair count values | 12 months
  The degree of improvement in hair quality and quantity using trichoscopic analyses will be based on the following:
  * Terminal to Vellus Ratio
  * Average hairs per follicular unit
  * Average hair width (mm)
  * Inter-follicular mean distance (mm)
  * Improvement in scalp hair appearance (blinded reviewers)

CONTACTS AND LOCATIONS:
Locations (1):
- UnionDerm, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No